CLINICAL TRIAL: NCT04527835
Title: Presentation, Clinical Course and Patterns of Myocardial Damage Due to Viral Myocarditis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shery Refaat Asaad, principal investigator, Assiut University
Other Study IDs: Viral myocarditis
Record Dates: First submitted 2020-08-23; First posted 2020-08-27 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-08

CONDITIONS: Viral Myocarditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients suspected for viral myocarditis: All patients admitted with unexplained heart failure in the last 3 months will be investigated for viral myocarditis by the use of 12 lead ECG, echocardiography, Cardiac MRI , coronary angiography, Endomyocardial biopsy ( optional ), serological tests including ELIZA,Extraction of nucleic acid, Determination of viral genome by using PCR., Quantitative real-time PCR to assess viral load, Immunohistochemistry analysis of EMB.
  Interventions: Diagnostic Test: ELIZA, Extraction of nucleic acid ,Determination of viral genome by using PCR, Quantitative real-time PCR to assess viral load ,Immunohistochemistry analysis of EMB.

INTERVENTIONS:
Diagnostic Test: ELIZA, Extraction of nucleic acid ,Determination of viral genome by using PCR, Quantitative real-time PCR to assess viral load ,Immunohistochemistry analysis of EMB. — ELIZA, Extraction of nucleic acid ,Determination of viral genome by using PCR, Quantitative real-time PCR to assess viral load ,Immunohistochemistry analysis of EMB.

SUMMARY:
Presentation, Clinical Course and Patterns of Myocardial Damage due to Viral Myocarditis

DETAILED DESCRIPTION:
1. Determine the pattern of myocarditis in hospitalized patients with acute HF within the last 3 months.
2. Determine the pattern of broad spectrum cardiotropic viruses in patients with acute HF within the last 3 months. These viruses like enteroviruses, adenoviruses and parvo B19 virus, HBV, HCV and Covid 19 virus due to its increased prevelance nowadays.

ELIGIBILITY:
Inclusion Criteria: All patients admitted with symptoms , signs and echocardiographic finding suggesting myocarditis within 3 months from start of the symptoms. as acute heart failure, arrhythmias, typical chest pain with ST segment deviation in ECG . dilated cardiomyopathy associated with normal Coronary Angiography, history of upper respiratory tract infection within the last 3 months.

Exclusion Criteria:

1. Patients with significant coronary artery disease.
2. Patient with family history suggesting familial DCMP
3. Critically ill patients.
4. Patients who refuse to do coronary angiography . .
5. Patients with severe valvular heart disease.
6. Pregnant women
7. Patients with raised renal chemistry.
8. Echocardiographic finding showing LVEDD more than 6.5cm

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients complained of symptoms of moderate to severe heart disease including atypical chest pain, fatigue, reduced physical capacity, recently occurring cardiac arrhythmia, and/or dyspnea on exertion suggesting myocardial inflammation.
Sampling Method: Probability Sample
Enrollment: 18 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Determine the pattern of myocarditis in hospitalized patients with acute HF within the last 3 months | 6 months
  All patients admitted with symptoms , signs and echocardiographic finding suggesting myocarditis within 3 months from start of the symptoms. as acute heart failure, arrhythmias, typical chest pain with ST segment deviation in ECG . dilated cardiomyopathy associated with normal Coronary Angiography, history of upper respiratory tract infection within the last 3 months. All will be investigated for determine the pattern of viral myocarditis in those patients

SECONDARY OUTCOMES:
determination of the caustive organism | 6 months
  1. Determine the pattern of broad spectrum cardiotropic viruses in patients with acute HF within the last 3 months. These viruses like enteroviruses, adenoviruses and parvo B19 virus, HBV, HCV and Covid 19 virus due to its increased prevelance nowadays.

CONTACTS AND LOCATIONS:
Overall Officials: Ayman khairy, professor, Principal Investigator — Assiut University; Mohamed El Mokhtar, professor, Principal Investigator — Assiut University
Locations (1):
- Shery Refaat Asaad, Asyut, Egypt